CLINICAL TRIAL: NCT04169464
Title: The Renal Safety and Rates of Acute Kidney Injury (AKI) in Patients With Chronic HCV Undergoing Sofosbuvir Containing Direct Acting Antiviral Therapy
Brief Title: The Renal Safety in Patients With Chronic HCV Undergoing Sofosbuvir Containing Antiviral Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Dalia Kamal Zaafar Ali, Lecturer of Pharmacology and Toxicology, MTI University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID22218
Record Dates: First submitted 2019-11-17; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Egyptian Patients, HCV Treatment, Kidney Function
Keywords: HCV; DAAs; Egyptian patients; creatinine; insulin resistence; GFR

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group I (Other): A group of HCV infected patients treated with DAA therapy including Sofospovir
  Interventions: Drug: Sofosbuvir Oral Product

INTERVENTIONS:
Drug: Sofosbuvir Oral Product — to investigate the drug effect on renal function and insulin resistance

SUMMARY:
The aim of this study is to investigate the occurrence of AKI during antiviral therapy, when compared with baseline values in Egyptian patients.

In addition, the study aims to evaluate the change in insulin resistance value after treating patients from HCV.

DETAILED DESCRIPTION:
There are limited published data, currently, suggesting the risk of AKI during oral direct acting antiviral treatment. Most case reports and retrospective studies reported the presence of an intrinsic cause of renal injury, with most of the available biopsies showing acute tubular necrosis (ATN) and acute interstitial nephritis (AIN). Most of these patients had returned to baseline renal function on cessation of sofosbuvir combination therapy.

Recently it was found that a notable percentage of patients experienced a transient increase in creatinine during therapy, which could occasionally lead to a more than 50% decrease in patients' eGFR. Previous studies had also shown that the co-use of nonsteroidal anti-inflammatory drugs (NSAIDs) and recurrent ascites were at increased risk for AKI during sofosbuvir-based antiviral therapy (Brawn et al., 2018).

The primary endpoint of this study is to investigate the occurrence of AKI in Egyptian patients during antiviral therapy and to highlight its reasons and time of incidence in addition to the mechanism of this injury.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years Chronic infection with HCV GT 4 No prior HCV treatment experience

Exclusion Criteria:

* Co-infection with HBV or HIV, clinical evidence of ischemic heart disease, the presence of diabetic ketoacidosis, Patients admitted to the intensive care unit (ICU), or expected to undergo surgery during the study period, and Child Pough score C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
occurance of AKI during therapy | 3 months
  investigate the occurrence of AKI during antiviral therapy, defined as an increase of 0.3 mg/dL or 50% at least in serum creatinine level when compared with baseline values or more than a 25% reduction in (eGFR) when compared with baseline eGFR in Egyptian patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Zaafar, Phd, Principal Investigator — Lecturer of pharmacology and toxicology
Locations (1):
- Thabet Thabet hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD are accepted to be shared in some cases where patients code only used without individual name